CLINICAL TRIAL: NCT06884241
Title: Effects of a Probiotic Supplementation on Symptoms and Microbiome Characteristics in Patients With Non-celiac Gluten/Wheat Sensitivity. A Randomized Controlled Double-blind Trial.
Brief Title: Effects of a Probiotic Supplementation on Symptoms and Microbiome Characteristics in Patients With Non-celiac Gluten/Wheat Sensitivity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLUTEN_2024
Record Dates: First submitted 2025-03-07; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Gluten Sensitivity; Wheat Sensitivity
Keywords: gluten sensitivity; wheat sensitivity; probiotics; microbiome
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants in this arm received a supplementation of probiotics for 6 weeks.
  Interventions: Dietary Supplement: Probiotic supplementation
- Control arm (Placebo Comparator): Participants in this arm received placebo for 6 weeks. The placebo were identical in size, shape, color, and taste to the probiotic.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation — The intervention consists of a 6-week supplementation with a specific combination of probiotics: Lactiplantibacillus plantarum P17630 49x109, Lacticaseibacillus paracasei I1688 1x109, Ligilactobacillus salivarius I1794 25x106. All participants were given a gluten-free, low FODMAPs diet. After 4 weeks (T1), foods containing gluten were reintroduced in the diet of all participants (at least 6 g/day of gluten), while the reduced FODMAP content was maintained
  Arms: Intervention arm
Other: Placebo — The participants received placebo for 6 weeks. Placebo was identical in appearance, texture, taste, and packaging to the probiotic treatment. All participants were given a gluten-free, low FODMAPs diet.
  After 4 weeks (T1), foods containing gluten were reintroduced in the diet of all participants (at least 6 g/day of gluten), while the reduced FODMAP content was maintained
  Arms: Control arm

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled clinical trial is to investigate the effects of probiotics on symptoms and gut microbiota composition following gluten reintroduction.

The study included adults diagnosed with NCWS. Participants received a 6-week intervention with either probiotics or a placebo. For the first 4 weeks, all participants followed a gluten-free, low-FODMAP diet, after which gluten was reintroduced.

Gastrointestinal symptoms (using the modified Gastrointestinal Symptom Rating Scale (GSRS)) and fecal samples were collected at baseline (T0), after 4 weeks (T1), and after 6 weeks (T2). Gut microbiome composition was assessed through whole-shotgun metagenomic sequencing and fecal volatile organic compounds (VOCs) were analyzed using gas chromatography-mass spectrometry (GC-MS).

DETAILED DESCRIPTION:
Non-Celiac Gluten Sensitivity (NCGS), or Non-Celiac Wheat Sensitivity (NCWS), is a condition characterized by the onset of gastrointestinal and systemic symptoms following the consumption of gluten-containing foods, without the presence of celiac disease or wheat allergy.

The aim of the present randomized, double-blind controlled trial is to explore probiotics as a potential therapeutic option to alleviate symptoms and improve gut microbiome composition.

Participants Eligible participants were adults aged 18 or older with NCGWS, confirmed by a positive response to the double-blind placebo-controlled (DBPC) cross-over gluten challenge test. Those with conditions like Crohn's disease, wheat allergy, IBS, gastrointestinal issues, infections, psychiatric disorders, or those on specific medications, as well as pregnant or breastfeeding individuals, were excluded.

Intervention Participants were randomized to receive for 6 weeks 2 sachets of probiotics (Lactiplantibacillus plantarum P17630 49x109, Lacticaseibacillus paracasei I1688 1x109, Ligilactobacillus salivarius I1794 25x106) (experimental arm) or 2 sachets of placebo (control arm). All participants a gluten-free and low FODMAPs diet. After 4 weeks, foods containing gluten were reintroduced in the diet of all participants (at least 6 g/day of gluten).

The investigators and the participants were blinded to the procedure. The probiotic and placebo sachets were identical and in identical packaging.

Measurements

At baseline (T0), after 4 weeks (T1, end of gluten-free diet), and after 6 weeks (T2, study-end), participants were submitted to the following measurements:

* modified GSRS questionnaire
* collection of a fecal sample for gut microbiota determination. At T1 and T2, volatile organic fractions of stool samples were assessed and whole shotgun metagenomics were performed.

ELIGIBILITY:
Inclusion criteria:

* age≥18 years
* NCGWS demonstrated by the following self-reported conditions i) intestinal and extra intestinal symptoms associated within hours or days after the ingestion of gluten-containing food, ii) a clear benefit while on a gluten-free diet, iii) relapse of symptoms with the ingestion of gluten-containing foods, iv) a positive response to the double-blind placebo-controlled (DBPC) cross-over gluten challenge test, as previously described.

Exclusion criteria:

* presence of Crohn disease (CD), wheat allergy (WA), irritable bowel syndrome (IBS), and other gastrointestinal diseases, H. Pylori infection, lactose intolerance, history of gastrointestinal surgery, liver/pancreatic diseases, active or recent infection diseases, known psychiatric diseases, any systemic diseases
* pregnancy or breastfeeding
* active use of antibiotics, pre-probiotics, immunosuppressive drugs, non-steroidal anti-inflammatory drugs, or corticosteroids,
* inability to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Symptoms Following Gluten Reintroduction | Symptoms were assessed at baseline (T0), after 4 weeks of a gluten-free diet (T1), and after 2 weeks of gluten reintroduction (T2).
  The primary outcome was evaluating between-group differences in symptoms reported by participants after gluten reintroduction, as measured by the modified Gastrointestinal Symptom Rating Scale (GSRS), according to the Salerno Experts criteria. Participants were defined as "tolerant" to the gluten-containing diet if their total GSRS scores did not change or reduced 2 weeks after the gluten introduction (T2)

SECONDARY OUTCOMES:
Gut microbiome composition after probiotic supplementation | Gut microbiome was analyzed at baseline (T0), after 4 weeks of a gluten-free diet (T1), and after 2 weeks of gluten reintroduction (T2).
  The assessment of gut microbiome composition after probiotic supplementation. Gut microbiome composition was assessed through whole-shotgun metagenomic sequencing.
Fecal volatilome after probiotic supplementation | Volatilome was analyzed at baseline and after 4 weeks of a gluten-free diet (T1), and after 2 weeks of gluten reintroduction (T2).
  The assessment of volatilome after probiotic supplementation by gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, Associate Professor, MD, Principal Investigator — University of Torino; Ilario Ferrocino, Professor, Study Director — University of Turin, Italy
Locations (1):
- AOU Città della Salute e della Scienza di Torino, University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No